CLINICAL TRIAL: NCT00083824
Title: Estrogen, HDL, and Coronary Heart Disease in Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stefania lamon-Fava, Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1253; R01HL070081 (NIH)
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Coronary Artery Disease | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone Acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Estrogens, Conjugated (USP) (Experimental): Conjugated Equine Estrogen 0.625 mg/day for 3 years, drug
  Interventions: Drug: Estrogens, Conjugated (USP)
- Medroxyprogesterone 17-acetate (Experimental): Conjugated Equine Estrogen 0.625 mg/day plus Medroxyprogesterone Acetate 2.5 mg/day
  Interventions: Drug: Estrogens, Conjugated (USP); Drug: Medroxyprogesterone 17-Acetate

INTERVENTIONS:
Drug: Estrogens, Conjugated (USP) — 0.625 mg/day QID for 3 years
  Other Names: Premarin
  Arms: Estrogens, Conjugated (USP); Medroxyprogesterone 17-acetate
Drug: Medroxyprogesterone 17-Acetate — 2.5 mg/day QID for 3 years
  Other Names: Provera
  Arms: Medroxyprogesterone 17-acetate
Drug: Placebo — 2 pills/day QID for 3 years
  Other Names: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
To clarify the effects of estrogen, with or without progestin, on high density lipoprotein (HDL) in postmenopausal women.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) is the leading cause of death and disability in postmenopausal women in the United States. Low plasma levels of high-density lipoprotein cholesterol (HDL-C) are a well-established risk factor for CHD. Elevated plasma triglyceride (TG) levels are also a risk factor for CHD in women. HDL particles are heterogeneous in composition (containing apo A-I only, LpAI, or apo A-I and apo A-II, LpAIAII) and charge and size (preBeta1, preBeta2, alpha1-3, preAlpha1-4). Different HDL subpopulations have different physiological functions and therefore may vary in their anti-atherogenic potential. Changes in alpha1 HDL subpopulations are a predictor of coronary disease progression in men. Hormonal replacement therapy (HRT) increases plasma levels of HDL-C, but has adverse effects on TG and C-reactive protein (CRP) levels. While observational studies had indicated a protective role of HRT in CHD, recent intervention studies have shown no CHD protection with the use of HRT. Our preliminary data indicate that there is a large inter-individual variability in HDL subpopulations and TG-rich lipoprotein remnants response to HRT.

The study uses the Estrogen Replacement and Atherosclerosis (ERA) trial which offers a unique opportunity to clarify the effects of estrogen with or without progestin on HDL and its subpopulation and TG-rich particles, and the effect of genetic polymorphisms on the response of these parameters to HRT. In addition, the ERA study will allow testing of the hypothesis that HRT may be of benefit to those postmenopausal women who experience large increases in HDL subpopulations (regardless of their overall effect on HDL cholesterol), without significant changes in TG levels. In addition, by looking at the TG and remnants of TG-rich lipoproteins, this study will enable a dissection of the beneficial and the adverse effects of HRT. The ERA population consists of 309 postmenopausal women who have established CHD and have participated in a randomized, placebo controlled, double-blind study of the effects of placebo (n-105), estrogen (n=100), and estrogen plus progestin (n=104) on the progression of coronary atherosclerosis, as assessed by quantitative coronary angiography. The trial showed no difference in coronary atherosclerosis progression across treatment groups after a mean follow-up of 3.2 years.

DESIGN NARRATIVE:

The study will clarify the effects of estrogen, with or without progestin, on HDL and its subpopulations and on lipoprotein remnants. It will also examine the impact of changes in HDL subpopulations and in lipoprotein remnants during HRT on progression of coronary atherosclerosis. These studies will be conducted in participants in the Estrogen Replacement and Atherosclerosis (ERA) trial, a randomized, placebo-controlled study of HRT and progression of atherosclerosis in postmenopausal women with CHD (n=309), in whom baseline and follow-up angiographic measurements of coronary artery diameter have been obtained. The following HDL parameters will be measured: preBeta1, preBeta2, alpha1-3, preAlpha1-4 HDL subpopulations by 2dGE, LpAI and LpAIAII in plasma and apo C-III in HDL and total plasma by immuno-electrophoresis, lipoprotein remnants by an immunoseparation method, and polymorphisms at gene loci involved in HDL metabolism (lipoprotein lipase, hepatic lipase, cholesteryl ester transfer protein, scavenger receptor B1, and ATPA1 receptor). Hypotheses tested are: 1) these HDL parameters and lipoprotein remnants will be significantly associated with severity of CHD at baseline; and 2) HRT-related changes in these parameters will predict coronary atherosclerosis progression in the ERA participants.

ELIGIBILITY:
Inclusion criteria:

age >55 years without natural menses for at least 5 years or a serum FSH levels >40 IU/L without natural menses for at least 1 y or bilateral oophorectomy documented coronary artery disease

Exclusion criteria:

history of breast or endometrial carcinoma history of deep-vein thrombosis or pulmonary embolism previous or planned coronary bypass gallstones fasting TG levels >400 mg/dl uncontrolled diabetes uncontrolled hypertension serum creatinine >2 mg/dl a >70% stenosis of the left main coronary artery.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2004-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
HDL subpopulation distribution and composition | 1 year
  To assess the effect of hormonal replacement therapy on HDL subpopulation profile and HDL composition in postmenopausal women with established CHD

SECONDARY OUTCOMES:
Remnant lipoprotein cholesterol | 1 year
  To assess the effect of hormonal replacement therapy on remnant lipoprotein cholesterol levels in postmenopausal women with established CHD

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Lamon-Fava, Principal Investigator — Tufts University; David M Herrington, MD, Study Director — Wake Forest University
Locations (1):
- HNRCA at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Herrington DM, Reboussin DM, Brosnihan KB, Sharp PC, Shumaker SA, Snyder TE, Furberg CD, Kowalchuk GJ, Stuckey TD, Rogers WJ, Givens DH, Waters D. Effects of estrogen replacement on the progression of coronary-artery atherosclerosis. N Engl J Med. 2000 Aug 24;343(8):522-9. doi: 10.1056/NEJM200008243430801. PMID 10954759
- [Result] Lamon-Fava S, Herrington DM, Reboussin DM, Sherman M, Horvath K, Schaefer EJ, Asztalos BF. Changes in remnant and high-density lipoproteins associated with hormone therapy and progression of coronary artery disease in postmenopausal women. Atherosclerosis. 2009 Jul;205(1):325-30. doi: 10.1016/j.atherosclerosis.2008.12.020. Epub 2008 Dec 24. PMID 19155011
- [Result] Lamon-Fava S, Herrington DM, Reboussin DM, Sherman M, Horvath KV, Cupples LA, White C, Demissie S, Schaefer EJ, Asztalos BF. Plasma levels of HDL subpopulations and remnant lipoproteins predict the extent of angiographically-defined coronary artery disease in postmenopausal women. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):575-9. doi: 10.1161/ATVBAHA.107.157123. Epub 2008 Jan 3. PMID 18174456
- [Result] Lamon-Fava S, Asztalos BF, Howard TD, Reboussin DM, Horvath KV, Schaefer EJ, Herrington DM. Association of polymorphisms in genes involved in lipoprotein metabolism with plasma concentrations of remnant lipoproteins and HDL subpopulations before and after hormone therapy in postmenopausal women. Clin Endocrinol (Oxf). 2010 Feb;72(2):169-75. doi: 10.1111/j.1365-2265.2009.03644.x. Epub 2009 May 29. PMID 19489872
- [Result] Lamon-Fava S, Herrington DM, Horvath KV, Schaefer EJ, Asztalos BF. Effect of hormone replacement therapy on plasma lipoprotein levels and coronary atherosclerosis progression in postmenopausal women according to type 2 diabetes mellitus status. Metabolism. 2010 Dec;59(12):1794-800. doi: 10.1016/j.metabol.2010.05.012. Epub 2010 Jun 26. PMID 20580029